CLINICAL TRIAL: NCT07407569
Title: Developing a First-void Urine-based Infection Model to Study HPV-specific Antibody-virion Interaction Before and After Vaccination With the Gardasil-9 HPV Vaccine - a Non-randomized Open-label Study.
Brief Title: Developing a First-void Urine-based Infection Model to Study HPV-specific Antibody-virion Interaction Before and After HPV Vaccination
Acronym: URVIVE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Hospital, Antwerp (Other); University Hospital, Ghent (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Wiebren Tjalma, Prof. Dr. Wiebren A.A Tjalma, Universiteit Antwerpen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025-522053-18-00; 2025-522053-18-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-22; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Human Papilloma Virus Infection Type 16
Keywords: HPV-specific antibodies; Gardasil 9; Vaccination; Self-sampling; First-void urine
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine nonavalent; Clinical Protocols

STUDY DESIGN:
Intervention Model Description: Exploratory, off-label use of authorized IMP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gardasil 9 Vaccination (Experimental): Single arm
  Interventions: Biological: Gardasil 9 (2 dose regimen)

INTERVENTIONS:
Biological: Gardasil 9 (2 dose regimen) — All subjects will be administered a 0.5 mL dose of the vaccine as an intramuscular injection in the deltoid following a two-dose schedule (0 months and 6 months).
  The Gardasil 9 vaccine is authorized and indicated for active immunization in individuals from the age of 9 years for the prevention of premalignant lesions and cancers aeecting the cervix, vulva, vagina and anus and genital warts caused by HPV types.

SUMMARY:
The current study is an open-label, non-randomized, longitudinal exploratory trial using the licensed Gardasil 9 (9vHPV) vaccine in an off-label context to investigate biological and immunological outcomes in human papillomavirus type 16 (HPV16) positive women. Two doses of the licensed Gardasil 9 vaccine will be administered to approximately 50 women between 18 and 45 years old, who test positive for HPV16 DNA at baseline using a type-specific quantitative PCR assay, but have no presence of apparent anogenital lesions and are thus not referred for treatment or intervention at the time of inclusion.

The primary objective of this study is to demonstrate that vaccination with a two-dose regimen of the 9vHPV vaccine reduces the viral infectivity of particles in the female genital tract of HPV16-positive women, by using first-void urine samples. The secondary objectives are to follow up HPV type-specific antibody responses in these first-void urine samples after natural infection and vaccination after one or two doses of the 9vHPV vaccine and to compare these with the responses in serum, and to monitor HPV infections in first-void urine over time.

Candidates will be selected for participation based on the result of their HPV DNA test performed on a sample collected during routine screening or symptomatic (opportunistic) testing in one of the following centers:

* The University Hospital of Antwerp (UZA).
* The University Hospital of Leuven (UZ Leuven).
* Ghent University Hospital (UZ Gent).

Women are followed for up to 24 months, in which first-void urine and serum samples will be collected at different timepoints.

The following laboratory procedures will be applied to reach study objectives

* Assessment of HPV DNA positivity: HPV genotyping in first-void urine samples.
* Assessment of HPV infectivity: Detection of HPV16 E1^E4 spliced mRNA in HaCaT keratinocytes after infection with virions from first-void urine samples.
* Assessment of HPV immunogenicity: Detection of HPV-specific antibodies in first-void urine and serum samples.

ELIGIBILITY:
Candidates are eligible for inclusion in the study if they:

* Are females between 18 and 45 years old (including both limits) at the time of signing the informed consent form.
* Have tested positive for HPV16 DNA (single or co-infection) but have no presence of apparent anogenital lesions and are thus not referred for treatment or intervention at the time of inclusion or within the last twelve months before inclusion.
* Did not receive prior vaccination with a prophylactic HPV vaccine.
* Are able to understand the information brochure and what the study is about.
* Are willing to give informed consent to the study team to access their medical records, including details on their HPV vaccination schedule and cervical cancer screening results (smears, HPV tests, colposcopy, biopsy).

Candidates must be excluded from the study if they:

* Are previously (completely or partially) vaccinated against HPV or have planned administration of another HPV vaccine during the study.
* Are pregnant at the time of signing informed consent or are planning to become pregnant within the full duration of the study. Participants must use an effective method of contraception throughout the entire study. Acceptable methods include combined hormonal contraception (oral, vaginal ring, transdermal patch), progestogen-only contraception (oral, injectable, implantable), intrauterine device (IUD)/intrauterine system (IUS), condom, vasectomized male partner, or (periodic) abstinence. Lactating women may be included.
* Have had full hysterectomy.
* Have had any anogenital lesion treated in the last twelve months before participating in the study.
* Have invasive cancer (except basocellular carcinoma) or other immunocompromising conditions as described as high-risk in the latest scientific guidelines from Sciensano.
* Use immunosuppressive therapy for inflammatory bowel disease, rheumatological disorders, neuromyelitis optica, sarcoidosis, adenocarcinoma in situ, or use of local anogenital corticosteroids.
* Have used any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planning to use during the study period.
* Have received immunoglobulin or blood-derived products in the three months prior to the first study vaccination (Month 0), or are expected to require immunoglobulin or blood-derived products from Month 1 until Month 7 of the study.
* Receive any vaccine not foreseen in the study protocol administered in the period beginning 30 days preceding each dose of the study vaccine and ending one month (minimum 30 days) after each dose of the study vaccine.
* Have known allergy or history of any reaction or hypersensitivity likely to be exacerbated by any component of the Gardasil 9 vaccine or known history of severe allergic reaction to other vaccines (e.g. anaphylaxis).
* Are concurrently enrolled in another clinical study of investigational agents.
* Have acute disease or contraindications for vaccination at the time of enrolment. Acute disease is defined as the presence of moderate or severe illness with or without fever. Enrolment will be deferred until the condition is resolved. All vaccines can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness, i.e. oral/axillary temperature >37.5 °C.
* Have a history or current evidence of any condition or abnormality that might confound the results of the study or is not in the best interest of the individual to participate, in the opinion of the investigator.
* Are, as determined by the investigator, unlikely to adhere to the study procedures, keep appointments, or are planning to relocate from the area prior to completion of the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Detection of HPV16 E1^E4 spliced mRNA in an in vitro infection model using first-void urine samples | 24 months
  Presence and relative expression level of HPV16 E1^E4 spliced mRNA in HaCaT keratinocytes following in vitro infection with HPV virions isolated from first-void urine samples collected before and after administration of two doses of the Gardasil 9 vaccine.

SECONDARY OUTCOMES:
Detection of HPV type-specific antibodies in first-void urine and serum samples | 24 months
  Presence and level of HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 type-specific antibodies in paired first-void urine and serum samples collected before and after administration of one or two doses of the Gardasil 9 vaccine.
Detection of HPV DNA in first-void urine samples | 24 months
  Presence of HPV DNA for genotypes 6, 11, 16, 18, 26, 31, 33, 35, 39, 40, 42, 43, 44, 45, 51, 52, 53, 54, 56, 58, 59, 61, 66, 68, 69, 70, 73, and 82 in first-void urine samples collected during follow-up.

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - Antwerp University Hospital, Antwerp, Wilrijk
  - University Hospital Ghent, Ghent
  - University Hospital Leuven, Leuven